CLINICAL TRIAL: NCT04708210
Title: An Open-label, Multicenter, Phase Ia/Ib Study to Evaluate the Safety, Tolerance and Preliminary Efficacy of IBI319 in Patients With Advanced Malignant Tumors
Brief Title: Study of the Efficacy and Safety of IBI319 in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI319A101
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ia Dose-Escalation Stage: IBI319 (Experimental)
  Interventions: Drug: IBI319

INTERVENTIONS:
Drug: IBI319 — Iv infusion day 1 of every 14 or 21 days in Phase Ia until disease progression or loss of clinical benefit.

SUMMARY:
An open-label, multicenter, phase Ia/Ib study to evaluate the safety, tolerance and preliminary efficacy of IBI319 in patients with advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Patients with advanced solid tumors or hematological malignancies who had failed standard treatment.
3. Male or female subjects ≥18 years and ≤75 years.
4. At least one measurable lesion (per RECIST version 1.1) in solid tumor patients and at least one measurable and hyper metabolic in 18F-FDG lesion (per Lugano2014) in lymphoma patients
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
6. Subjects with life expectancy of ≥ 12 weeks.
7. Subjects must have adequate organ function (liver, kidney function and hematopoietic function tests) prior IBI319 administration

   1. Absolute neutrophil count (ANC) ≥1.5 x10^9/L
   2. Platelet count ≥ 100 x 10^9/L
   3. Hemoglobin ≥ 9 g / dL (whole blood or component transfusion within 7 days before 1st dose of study drug is prohibited)
   4. Renal function tests: an estimated glomerular filtration rate (eGFR) ≥ 50 mL/min
   5. Liver function tests alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN, for patients with known liver cancer or liver metastases, AST and ALT ≤ 5 x ULN
   6. Total bilirubin (TBil) ≤1.5 x ULN; If Gilbert's Syndrome may have Bilirubin> 2 x ULN
   7. Coagulation tests: APTT ≤ 1.5 x ULN and INR ≤1.5 x ULN
8. Subjects (males and females) of childbearing potential should be willing to use reliable contraception methods that are deemed effective by the investigator from visit 1 through 180 days following the last dose of study drug.

Exclusion Criteria:

1. Legal incapacity or limited legal capacity.
2. Pregnancy, lactation, breastfeeding.
3. Prior treatment with an anti-CD137, anti-Programmed Death Receptor (PD)-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-Cell Lymphoma-4 Antigen (CTLA-4) antibody, or any other antibody or drug (except for Ib cohort A and B).
4. NSCLC patients with EGFR mutations or ALK gene rearrangements.
5. Colorectal cancer patients with KRAS mutation / BRAF mutation / HER2 overexpression.
6. Concurrent anticancer treatment or use of other investigational product within 4 weeks before start of trial treatment; major surgery within 4 weeks before start of trial treatment (excluding prior diagnostic biopsy).
7. Failure to recover from adverse events from the most recent anti-tumor treatment to CTCAE ≤ grade 1 or baseline with the exception of alopecia.
8. Acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
9. Subjects with CNS metastasis unless they are asymptomatic or adequately treated with radiotherapy and/or surgery and subjects are neurologically stable with minimal residual symptoms/signs.
10. Any other serious underlying medical (e.g., uncontrolled hypertension, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, other serious cardiac conditions not listed in exclusion criteria), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Number of patients with DLT, AE, treatment-related AE (TRAE), immune-related AEs (irAE), AE of special interest (AESI), serious adverse event (SAE), discontinuation of study drug due to AE, dose-limiting toxicity (DLT) assessed by CTCAE v5.0 | up to 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) based on RECIST v1.1 criteria and Lugano 2014 criteria. | up to 2 years
Progression-free survival (PFS) based on RECIST v1.1 criteria and Lugano 2014 criteria | up to 2 years
Overall Survival (OS) based on RECIST v1.1 criteria and Lugano 2014 criteria | up to 2 years
Time To Response(TTR) based on RECIST v1.1 criteria and Lugano 2014 criteria | up to 2 years
Duration of Response(DOR) based on RECIST v1.1 criteria and Lugano 2014 criteria | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, China